CLINICAL TRIAL: NCT01454011
Title: Phase 4 Study That Compares the High Density Lipoprotein Cholesterol (HDL) Cholesterol Subgroups of the Patients With Congenital Hypogonadotrophic Hypogonadism With That of the Healthy Control Subjects, and Investigates the Effect of Testosterone Treatment on HDL Subgroups.
Brief Title: The Effect of Testosterone Replacement on the High Density Lipoprotein Cholesterol Subgroups
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Associate Professor, Gulhane School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSM-012011
Record Dates: First submitted 2011-10-12; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Secondary Hypogonadism
Keywords: hypogonadism; testosterone; HDL cholesterol subgroups; hsCRP; HOMA-IR
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate; Injections; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone 250mg injection, (Active Comparator)
  Interventions: Drug: Testosteron 250mg injection
- Testosterone transdermal application (Active Comparator)
  Interventions: Drug: Testosterone 50mg transdermal application

INTERVENTIONS:
Drug: Testosteron 250mg injection — The combination of 4 different testosterone esthers (30 mg testosterone propionate, 60 mg testosterone phenylpropionate, 60 mg testosterone isocaproate and 100 mg testosterone decanoate) injected in 3 weeks intervals.
  Other Names: Sustanon 250 mg ampule
  Arms: Testosterone 250mg injection,
Drug: Testosterone 50mg transdermal application — Application of testosterone 50mg transdermal gel in every night
  Other Names: Testogel 50mg transdermal gel
  Arms: Testosterone transdermal application

SUMMARY:
The study is designed to answer the following questions:

1. Is there any difference between the compositions of the HDL cholesterol subpopulations of patients with hypogonadism and the healthy controls.
2. What is the effect of testosterone replacement therapy on the distributions of HDL subgroups.
3. Is there any difference between the effects of the two different testosteron replacement regiments

DETAILED DESCRIPTION:
This study has two designs:

1. The case control design to search for the difference between the HDL subgroups and the other metabolic parameters between the healthy subjects and the patients with hypogonadism
2. The follow-up study to search for the effects of two different testosterone replacement regiments.

ELIGIBILITY:
Inclusion Criteria:

* Congenital hypogonadotrophic hypogonadism,
* Male sex

Exclusion Criteria:

* Previous history of androgen replacement,
* any chronic disorder

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Changes in the HDL cholesterol levels and the HDL subgroups | 6 months
  The HDL subfractions were measured by polyethylene glycol (PEG) precipitation technique. Two different reagents were prepared in different PEG concentrations and pH values. The supernatant of the solution precipitated with reagent A contained total HDL cholesterol while the supernatant of the solution precipitated with reagent B, contained only the HDL3 subclass. The cholesterol was then quantified by enzymatic with CHOD-PAP reagent (Olympus Diagnostics GmbH, Hamburg, Germany). HDL2 cholesterol was measured by calculating the difference between total HDL and the HDL3 subclass.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)